CLINICAL TRIAL: NCT03482258
Title: The Effect of Prebiotic Galacto-oligosaccharide on Stress Related Eating Behaviours and Mood.
Brief Title: The Gut Microbiota in Stress, Mood and Eating Behaviours.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roehampton (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Ellie Haydon-Islam, PhD student, University of Roehampton
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 08459942
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Eating Behavior; Stress; Mood
Keywords: Stress; Galactooligosaccharide; Prebiotic; Early life stress; Emotional eating; Gut microbiota; Short-chain fatty acids; Serotonin; Cortisol
MeSH Terms: conditions — Feeding Behavior; Stress, Psychological; Emotional Eating | interventions — Prebiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Blinding of supplements will be conducted by Frieslandcampina who are providing both prebiotic and maltodextrin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Prebiotic (Experimental): 3 week daily dose of Vivinal-GOS (galacto-oligosaccharide)
  Interventions: Dietary Supplement: Prebiotic
- Placebo (Placebo Comparator): 3 week daily dose of Maltodextrin
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Prebiotic — A daily dose for 3 weeks -14.5g per day in powder form dissolved in 200ml water. This equates to 10g GOS (VGOS is primarily 69% GOS, 23% Lactose).
  Other Names: Vivinal-GOS
  Arms: Treatment Prebiotic
Dietary Supplement: Maltodextrin — A daily dose for 3 weeks -14.5g per day in powder form dissolved in 200ml water. This will be matched to VGOS for lactose (3.3g per dose of maltodextrin will be lactose).
  Arms: Placebo

SUMMARY:
Diet has a considerable influence on microbiota composition and the intake of either prebiotics (microbiota-specific food or probiotics (live microbiota species) has been shown to induce positive effects in both anxiety and depression. At present there are few studies exploring stress-related conditions such as emotional/comfort eating behaviours, particularly in individuals who have experienced early life stress and/or find stress difficult to deal with in regards to gut microbiome composition and subsequent behavioural outcomes. Early life stress has been linked to the development of bulimia nervosa and anorexia nervosa in adolescence and adulthood and since the gut microbiota has been proposed as having a causal role in the aetiology and/or maintenance of disordered eating, an empirical question is whether the microbiota may mediate the relation between stress and disordered eating. This is an investigation into the effects of chronic daily consumption of a prebiotic on stress-related eating and mood.

DETAILED DESCRIPTION:
Following an initial screening session based on inclusion/exclusion criteria, participants will be randomly allocated into either the treatment or placebo group and provided with three weeks worth of Vivinal-GOS or maltodextrin in powder form (sachets). There will be four clinical visits as detailed below:

1. Training on how to complete food diaries and collect saliva samples for cortisol awakening response measurements
2. Cognitive (Affective GoNoGo and Emotion Recognition Task) and biologic measurements (blood,faecal). This also includes a stress inducing task (Fake Speech Task).Provided with supplement and invited to next session in three weeks' time.
3. Cognitive (Affective GoNoGo and Emotion Recognition Task) and biologic measurements (blood,faecal). This also includes a stress inducing task (Fake Speech Task).
4. (one week after last visit) collection of final faecal sample

ELIGIBILITY:
Inclusion Criteria:

* A positive or negative screen for exposure to adverse childhood experiences
* A positive or negative screen for stress/emotional related eating behaviours
* Written informed consent

Exclusion Criteria:

* Antibiotic, prebiotic or probiotic use in past three months
* Pre-existing gastrointestinal disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Gut microbiota composition | 4 weeks
  A comparison of the microbiota between individuals who are or are not prone to stress/emotional eating behaviours potentially due to early life stress, and whether treatment with a prebiotic (GOS) alters this.
  Metagenomic studies will be conducted to evidence base outcomes linked to changes in microbial population
  1HNMR profiling will be used to identify biochemical/ bioactive mechanisms for regulatory needs

SECONDARY OUTCOMES:
Negative affect | 4 weeks
  To observe whether treatment with GOS moderates negative affect using cognitive tasks (Affective GoNoGo and Emotion Recognition test).
Gut Brain Axis | 4 weeks
  To gain further understanding of the mechanisms of the GBA by examining blood and/or faecal levels of SCFAs and TRP, in relation to behavioural outcomes and microbiota populations.
  SCFAs in serum will be measured via blood samples (ratio of acetate, propionate and butyrate) Levels of serum propionate in relation to satiety- plasma concentrations of PYY and GLP-1
Eating behaviour | 4 weeks
  To observe whether participants engage stress related eating behaviours (over-eating, eating high energy foods) and if prebiotics negate these behaviours.
  This will be measured via a exposure to a stressful situation (fake speech task) and subsequent food consumption (a meal will provided).
Stress response | 4 weeks
  To observe whether treatment with GOS moderates the stress response
  Cortisol awakening response will be measured via saliva samples.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Gibson, Study Director — University of Roehampton
Locations (1):
- University of Roehampton, London, United Kingdom